CLINICAL TRIAL: NCT06930144
Title: Immunomodulatory and Therapeutic Efficacy of 5-methyltetrahydrofolate Supplementation on Autoimmune Status in Type 1 Diabetes Mellitus
Brief Title: 5-MTHF Supplementation for Treatment of Type 1 Diabetes Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CZYZ-5MTHF-2025-IIT
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-MTHF supplementation group (Experimental): basic diabetes treatment combined with 5-MTHF (5-Methyltetrahydrofolate)
  Interventions: Drug: active folate
- placebo control group (Placebo Comparator): basic diabetes treatment combined with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: active folate — Daily oral intake of active folate 800ug combined with basic diabetic treatment
  Other Names: 5-Methyltetrahydrofolate
  Arms: 5-MTHF supplementation group
Drug: Placebo — take oral placebo daily combined with basic diabetic treatment
  Arms: placebo control group

SUMMARY:
This study aims to evaluate the improvement of autoimmune status in patients with Type 1 Diabetes (T1D) through supplementation with 5-Methyltetrahydrofolate, and to explore the safety and efficacy of this treatment. The research seeks to provide new methods for the treatment of T1D and offer innovative ideas for enhancing the quality of life of T1D patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with T1D based on the World Health Organization (WHO) classification criteria for disease diagnosis.
2. Aged 13-65 years, regardless of gender.
3. Duration of T1D ≤ 5 years.
4. Retained residual islet function, defined as fasting C-peptide > 0.1 nmol/L [0.30 ng/mL] or postprandial 2-hour C-peptide > 0.2 nmol/L [0.60 ng/mL].
5. Determined by the investigator to be capable and willing to: perform self-monitoring of blood glucose (SMBG); complete patient logs as required; receive diabetes education; and comply with the study treatment and visit schedule as per the protocol.

6) Signed informed consent form, with parental/guardian consent and signature required for pediatric/adolescent participants.

Exclusion Criteria:

1. Serum 5-methyltetrahydrofolate or folate levels exceeding the upper limit of the normal reference range.
2. Currently experiencing acute metabolic disorders, such as diabetic ketoacidosis or hyperosmolar hyperglycemic state.
3. Women who are breastfeeding, pregnant, or planning to become pregnant during the trial.
4. Received immunosuppressive or immunomodulatory therapy within the past year.
5. Comorbid with other autoimmune diseases, such as systemic lupus erythematosus.
6. Severe liver, kidney, gastrointestinal, hematologic, cerebral, or circulatory system diseases.
7. Psychiatric or neurological disorders leading to non-cooperation, non-adherence to medication, substance abuse, or other related issues.
8. Malignancy.
9. Recent surgery or significant stress.
10. Known hypersensitivity or allergic reaction to 5-methyltetrahydrofolate or its excipients.
11. Investigator's judgment of significant evidence of severe, active, or uncontrolled endocrine or autoimmune abnormalities.
12. Currently participating in another clinical trial.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Islet β cell function | From enrollment to 24 weeks of treatment
  Change in the area under curve (0-180min) of the serum C-peptide during the MMTT (Mixed Meal Tolerance Test) at 24 weeks of treatment.

SECONDARY OUTCOMES:
HbA1c | From enrollment to 24 weeks of treatment
  glycated hemoglobin (HbA1c) <7·0% or ≥ 1% reduction of HbA1c levels from baseline
lymphocyte subsets | From enrollment to 24 weeks of treatment
  change in lymphocytes subsets
islet autoantibodies | From enrollment to 24 weeks of treatment
  type and titer of islet autoantibodies
insulin dosage | 24 weeks of treatment
  change in insulin dosage at 24 weeks of treatment
cytokines | From enrollment to 24 weeks of treatment
  change in serum cytokines
CRP | From enrollment to 24 weeks of treatment
  change in C-reactive protein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vukotic R, Di Donato R, Roncarati G, Simoni P, Renzulli M, Gitto S, Schepis F, Villa E, Berzigotti A, Bosch J, Andreone P. 5-MTHF enhances the portal pressure reduction achieved with propranolol in patients with cirrhosis: A randomized placebo-controlled trial. J Hepatol. 2023 Oct;79(4):977-988. doi: 10.1016/j.jhep.2023.06.017. Epub 2023 Jul 22. PMID 37482222
- [Result] Verhaar MC, Wever RM, Kastelein JJ, van Dam T, Koomans HA, Rabelink TJ. 5-methyltetrahydrofolate, the active form of folic acid, restores endothelial function in familial hypercholesterolemia. Circulation. 1998 Jan 27;97(3):237-41. doi: 10.1161/01.cir.97.3.237. PMID 9462523
- [Result] Giammarco S, Chiusolo P, Maggi R, Rossi M, Minnella G, Metafuni E, D'Alo F, Sica S. MTHFR polymorphisms and vitamin B12 deficiency: correlation between mthfr polymorphisms and clinical and laboratory findings. Ann Hematol. 2024 Oct;103(10):3973-3977. doi: 10.1007/s00277-024-05937-z. Epub 2024 Aug 28. PMID 39196375